CLINICAL TRIAL: NCT03888131
Title: A 24-week, Double Blind, Double Dummy, Randomized, Multicentre, 2-arm Parallel Group, Active Controlled Clinical Trial of Fixed Combination of Beclometasone Dipropionate Plus Formoterol Fumarate Administered Via pMDI (CHF 1535) Versus the Fixed Combination of Budesonide Plus Formoterol Fumarate (Symbicort® Turbohaler®) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Foster® pMDI (CHF 1535) Versus Symbicort® Turbohaler in COPD Patient
Acronym: FORSYYN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCD-01535AC1-02
Record Dates: First submitted 2018-08-22; First posted 2019-03-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung functions; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHF 1535 100/6 µg pMDI (Experimental): 2 inhalations BID Total Daily Dose = 400/24µg
  Interventions: Drug: CHF 1535 100/6 µg pMDI plus Symbicort® Turbohaler® Placebo
- Symbicort® Turbohaler® (Active Comparator): 2 inhalations BID Total Daily Dose = 640/18µg
  Interventions: Drug: Symbicort® Turbohaler® plus CHF 1535 pMDI Placebo

INTERVENTIONS:
Drug: CHF 1535 100/6 µg pMDI plus Symbicort® Turbohaler® Placebo — Fixed combination of beclometasone dipropionate 100 µg plus formoterol fumarate 6 µg (BDP/FF)
  Arms: CHF 1535 100/6 µg pMDI
Drug: Symbicort® Turbohaler® plus CHF 1535 pMDI Placebo — Fixed combination of 160 µg budesonide + 4.5 µg formoterol fumarate (BUD/FF)
  Arms: Symbicort® Turbohaler®

SUMMARY:
The purpose of the study is to demonstrate the non-inferiority of CHF1535 pMDI versus Symbicort® Turbohaler® in terms of lung function parameters and patients reported outcomes and to assess its safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 40 years, Chinese ethnicity
* Patients with COPD diagnosed at least 12 months before the screening visit.
* A smoking history of at least 10 pack years
* Post-bronchodilator FEV1 < 50% of the predicted normal value
* Post-bronchodilator FEV1/FVC ratio < 0.7
* One exacerbation in the 12 months prior the screening visit

Exclusion Criteria:

* Patients requiring OCS/antibiotics/PDE inhibitors in the 4 weeks prior to screening
* COPD exacerbation requiring OCS/antibiotics or hospitalization during the run-in period
* Known respiratory disorders other than COPD
* Diagnosis of asthma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Demonstration of the non-inferiority of CHF 1535 pMDI versus Symbicort® Turbohaler® in terms of pulmonary function | At week 24
  Change from baseline in pre-dose morning First Expiratory Volume in 1 second (FEV1) in patients with Chronic Obstructive Pulmonary Disease (COPD)

SECONDARY OUTCOMES:
Effect of CHF 1535 on change from baseline pre-dose morning FEV1 | At week 4, week 12, week 18 and week 24
  FEV1 is the volume of air that can be forced out in one second after taking a deep breath. FEV1 will be measured via spirometer.
Effect of CHF 1535 on chnage from Baseline in pre-dose morning Force Vital Capacity (FVC) | At week 4, week 12, week 18 and week 24
  FVC is the volume of air expired after a maximum inspiration. FVC will be measured via spirometer.
Effect of CHF 1535 on change from baseline in the St. George's Respiratory Questionnaire (SGRQ) total scores and domains | At week 12, week 24
  The SGRQ is a well-established, self-completed tool to measure impact on overall health, daily life and perceived well-being in patients with obstructive airways disease. Score range from 0 to 100 with higher scores indicating more limitations.
Effect of CHF 1535 on change from baseline in COPD Assessment Test (CAT) | Over 28 weeks
  CAT is an easy questionnaire self-administered by patients. It was specifically designed to measure candidate items regarding daily symptoms, activity limitations and other manifestations of the COPD. It will be filled in at all clinical visits.
Effect of CHF 1535 on the rate of COPD exacerbations | Over 24 weeks of treatment
  The number of moderate and severe COPD exacerbations during the treatment period will be collected and analyzed.
  * Moderate exacerbations require treatment with systemic corticosteroids and/or antibiotics
  * Severe exacerbations require hospitalisation or result in death
Number of patients with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Over 29 weeks (from Visit 0 to Visit 6)
  An AE is "any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment".
  A SAE is defined as any untoward medical occurrence or effect that, at any dose may result in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Assessment of blood pressure | Over 28 weeks (from Visit 1 to Visit 6)
  Systolic and diastolic blood pressure will be measured at all clinical visits from Visit 1 after 10 minutes in seated resting position.
Number of subjects with abnormal Electrocardiogram (ECG) findings | At screening visit and week 24
  Twelve-lead ECG measurements will be obtained after the subject laid in a resting position for 10 minutes. ECG will be recorded in triplicate and evaluated at Visit 1 and Visit 6.
Number of subjects with abnormal Haematology parameters | At screening visit and week 24
  The following Haematology parameters will be assessed by a central laboratory: Red blood cells count (RBC), white blood cells count (WBC) and differential, total haemoglobin (Hb), hematocrit (Hct), platelets count (PLT).
Number of subjects with abnormal Blood Chemistry parameters | At screening visit and week 24
  The following Blood Chemistry parameters will be assessed by a central laboratory: creatinine, BUN, fasting serum glucose, aspartate aminotransferase (AST), alanine aminotransferase (ALT), Gamma-glutamyl transpeptidase (γ-GT), total bilirubin, alkaline phosphatase, sodium, potassium, calcium, and chloride electrolytes (Na, K, Ca, Cl), albumin.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Fuqiang WEN, M.D., Ph.D., Principal Investigator — West China Hospital
Locations (53):
- China (53):
  - Site 15604 - Anhui Provincial Hospital, Hefei, Anhui
  - Site 15635 - The Second Hospital of Anhui Medical Hospital, Hefei, Anhui
  - Site 15613 - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Site 15611 - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Site 15640 - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Site 15626 - Peking University Third Hospital, Beijing, Beijing Municipality
  - Site 15612 - Beijing Tong Ren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Site 15634 - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - Site 15616 - Chongqing Red Cross Hospital, People's Hospital of Jiangbei District, Chongqing, Chongqing Municipality
  - Site 15636 - Fujian Province Hospital, Fuzhou, Fujian
  - Site 15650 - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Site 15630 - Dongguan People's Hospital, Dongguan, Guangdong
  - Site 15607 - The First People's Hospital of Shunde, Foshan, Guangdong
  - Site 15619 - The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - Site 15608 - The First Affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Site 15646 - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Site 15651 - The Second Xiangya Hospital of Central South University, Guangzhou, Guangdong
  - Site 15614 - Guangzhou Panyu central hospital, Guangzhou, Guangdong
  - Site 15618 - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Site 15656 - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi Zhuang
  - Site 15637 - Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - Site 15623 - Haikou People's Hospital, Haikou, Hainan
  - Site 15645 - Hainan General Hospital, Haikou, Hainan
  - Site 15654 - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Site 15617 - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - Site 15622 - The Third Hospital of Changsha, Changsha, Hu'nan
  - Site 15647 - The Second hospital. University of South China, Hengyang, Hu'nan
  - Site 15653 - Xiangtan Central Hospital, Xiangtan, Hu'nan
  - Site 15603 - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Site 15657 - Zhong Da Hospital, Southeast University, Nanjing, Jiangsu
  - Site 15627 - Nanjing Medical University Affiliated 2nd Hospital, Nanjing, Jiangsu
  - Site 15621 - Wuxi People's Hospital, Wuxi, Jiangsu
  - Site 15632 - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Site 15659 - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Site 15658 - Jilin Province People's Hospital, Changchun, Jilin
  - Site 15643 - No.2 Hospital Affiliated to Jilin University, Changchun, Jilin
  - Site 15648 - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - Site 15649 - The 1st Affiliated Hospital of Shanxi Medical University, Taiyuan, Shan'xi
  - Site 15644 - Jinan Central Hospital, Jinan, Shandong
  - Site 15629 - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Site 15628 - Shanghai Xuhui Center Hospital, Shanghai, Shanghai Municipality
  - Site 15601 - Huadong Hospital Afflilliated to Fudan University, Shanghai, Shanghai Municipality
  - Site 15631 - Shanghai Yangpu District Centre Hospital, Shanghai, Shanghai Municipality
  - Site 15610 - Tong Ren Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Site 15606 - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Site 15625 - Central Hospital of Shanghai Minhang District, Shanghai, Shanghai Municipality
  - Site 15638 - Second Hospital of Shanxi Medical, Taiyuan, Shanxi
  - Site 15605 - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Site 15609 - Tianjin First Center Hospital, Tianjin, Tianjin Municipality
  - Site 15633 - Tianjin Haihe Hospital, Tianjin, Tianjin Municipality
  - Site 15602 - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Site 15642 - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Site 15639 -The second Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wen F, Wu Y, Xing C, Zhu Y, Chen Y, Mei X, Corradi M, Cappellini G, Calabro E, Amodio S, Zhu C, Galkin D. Beclometasone Dipropionate/Formoterol Fumarate is Similarly Effective to Budesonide/Formoterol Fumarate in Chinese Patients with COPD: The FORSYYN Double-Blind, Randomised Study. COPD. 2024 Dec;21(1):2425157. doi: 10.1080/15412555.2024.2425157. Epub 2024 Nov 11. PMID 39529298